CLINICAL TRIAL: NCT06301061
Title: Effectiveness of Focal Microvibration in the Management of Chronic Lumbosacral Radicular Pain: a Randomized Controlled Study
Brief Title: Focal Microvibration and Chronic Lumbosacral Radicular Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Maria Vargas, Prof, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PB001
Record Dates: First submitted 2024-02-15; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Pain, Chronic; Lumbosacral Radiculopathy; Radicular; Neuropathic
MeSH Terms: conditions — Chronic Pain; Radiculopathy | interventions — Gabapentin; Pregabalin; Duloxetine Hydrochloride; Amitriptyline; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients treated with Focal Microvibration (Experimental): Patients will be treated with focal microvibration through the application on the skin of four devices for 6 hours/day every day except thursady and Sunday.
  Interventions: Device: Equistasi®
- Patients treated with a Sham device (Sham Comparator): Patients will be treated with four sham device which will be attached on the skin for 6 hours/day every day except thursady and Sunday.
  Interventions: Device: Sham
- Patients treated with standard pharmacological approach (Active Comparator): Patients will be treated with standard pharmacological therapy
  Interventions: Drug: Gabapentin; Pregabalin; Duloxetine; Amitriptyline

INTERVENTIONS:
Device: Equistasi® — Four devices will be attached to the skin according the indication of the investigators for 6 hours/day every day except Thursday and Sunday
  Arms: Patients treated with Focal Microvibration
Device: Sham — Four devices similar to the active one but not able to deliver the microvibration will be applied to the patients
  Other Names: No active device
  Arms: Patients treated with a Sham device
Drug: Gabapentin; Pregabalin; Duloxetine; Amitriptyline — Patients will be treated with drugs (gabapentinoids, Serotonin-norepinephrine reuptake inhibitor, tricyclic antidepressants, opioids) according to guidelines.
  Other Names: Drugs for neuropathic pain
  Arms: Patients treated with standard pharmacological approach

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of focal microvibration on patients affected by chronic lumbosacral radicular pain. The main question[s] it aims to answer are:

* Can focal microvibration improve pain in this patient population?
* Can focal microvibration improve quality of life in these patients? Participants will attach to their skin four little devices (10x20x0,5mm) delivering focal microvibration in the painful area according to researchers indications for 6 hours/day every day except Thursday and Sunday.

Researchers will compare patients treated with focal microvibration to patients treated with a sham device and to patients treated with standard pharmacological therapy.

DETAILED DESCRIPTION:
This is the first randomized controlled study aiming to assess the potential use of focal microvibration for the management of chronic lumbosacral radicular pain which is the pain consequent to the compression of a spinal nerve root. Focal microvibration has been so far used to treat gait disorders and instability consequent to diseases such as Parkinson's disease, stroke, ataxia, multiple sclerosis with impressive results and no reported side effects. Our trial involves three arms: one arm treated with a device able to deliver focal microvibration, one arm treated with a sham device, and one arm treated with standard pharmacological therapy according to international guidelines. Patients with the active and with sham devices will attach them on their skin for 6 hours/day except on Thursday and Sunday: this application schedule with two days of treatment suspension has intended to avoid habituation to the sub-perception microvibration stimulation. The follow up will be 12 months and periodic visits will be performed after 7, 15 30, 45, 60, 90, 180, and 360 days of treatment. All the patients enrolled in the study will have access to rescue analgesic drugs such as paracetamol 1g and tramadol 100mg in case on excessive pain. Randomization will be performed by a computer-generated sequence. During the follow up visits, patients will be asked to fill questionnaires to explore and monitor pain intensity and pain interference in daily life: brief pain inventory (BPI) and Oswestry disability index (ODI)

ELIGIBILITY:
Inclusion Criteria:

* Pain duration≥6 months
* Magnetic resonance imaging (MRI) showing compression of lumbosacral nerve roots
* Neuropathic symptoms in the innervation territory of the compressed spinal nerve roots
* Monolateral pain
* Pain intensity: moderate-severe i.e. numeric rating scale (NRS)≥4.

Exclusion Criteria:

* Psychiatric patients
* Cancer patients
* Patients affected by disease characterized by spasticity or muscular stiffness:

Parkinson's disease, multiple sclerosis, stroke, spine injuries.

* Patients with spinal or dorsal root ganglion stimulators
* Patients undergone central of peripheral stimulation in the past 3 months
* Patients affected by fibromyalgia.
* Patients undergone central nervous system surgery
* Patients with reduced renal function eGFR≤60ml/min/1,73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 12 months
  Change in pain intensity with numeric rating scale (NRS): NRS ranges from 0 (no pain) to 10 (the the worst pain imaginable)

SECONDARY OUTCOMES:
Pain interference in daily life | 12 months
  Pain interference in patient daily life: mood, general activity, social relationship, work ability measured by Brief Pain Inventory (BPI). BPI is a 9 item self-administered questionnaire and every item score ranges from 0 to 10: a higher score indicates a worst outcome.
Disability | 12 months
  Disability related to pain severity measured by and Oswestry Disability Index (ODI). ODI score ranges from 0 to 100; a higher score on the ODI indicates a more severe disability caused by low back pain.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buonanno P, Iacovazzo C, Marra A, de Siena AU, Josu T, Zampi M, Sedda D, Servillo G, Vargas M. Potential Role of Focal Microvibration (Equistasi(R)) in the Management of Chronic Pain: A Pilot Study. Pain Ther. 2024 Feb;13(1):185-198. doi: 10.1007/s40122-023-00562-6. Epub 2023 Dec 6. PMID 38057548